CLINICAL TRIAL: NCT02288663
Title: Renal Function Assessment in the Elderly Using Plasma Creatinine Assay and Lean Body Mass Measurement
Acronym: FREAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5744
Record Dates: First submitted 2014-07-08; First posted 2014-11-11 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Renal Function
MeSH Terms: interventions — Albumins; Blood Specimen Collection; Urination; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Freage group (Other): only one group in this trial. All the participants will follow all the listed interventions.
  Interventions: Other: measurement of morphological parameters; Biological: a blood sample; Biological: albumin or blood in urine; Device: Dual X-ray absorptiometry (DXA); Device: Bioelectric Impedance Spectroscopy (BIS); Biological: 51Cr-EDTA plasma clearance

INTERVENTIONS:
Other: measurement of morphological parameters — measurement of morphological parameters : thigh perimeter, leg perimeter, arm perimeter.
Biological: a blood sample — One single blood sample to assay SCr (enzymatic), BUN (blood urea nitrogen), cystatin C, CRP, Na, K, Cl, albuminemia.
Biological: albumin or blood in urine — dipstick analysis for albumin or blood in urine
Device: Dual X-ray absorptiometry (DXA) — measurement of lean body mass by whole-body DXA
Device: Bioelectric Impedance Spectroscopy (BIS) — measurement of lean body mass by BIS
Biological: 51Cr-EDTA plasma clearance — measurement of 51Cr-EDTA plasma clearance to determine GFR

SUMMARY:
Glomerular filtration rate (GFR) is the recommended parameter to assess renal function. The reference technique to measure GFR (clearance of a glomerular agent) is not commonly used. Instead, estimations (eGFR) are routinely taken from serum creatinine (SCr) with several published formulae: Cockcroft and Gault, MDRD, CKD-EPI. Basically, all these formulae aim at predicting the endogenous creatinine production by morphological parameters (age, body weight...) However, in the elderly, muscular mass is extremely variable and sarcopenia is quite commonly encountered (frequently linked to Alzheimer disease). This is probably the main reason why the aforementioned formulae are not valid in this population: for a given renal function, a lower muscular mass induces a lower creatinine production and, henceforth, a lower SCr value, which gives an overestimation of eGFR.

Muscular mass is closely linked to lean body mass (LBM), which can be properly assessed by whole-body dual X-ray absorptiometry (DXA). Alternatively, Bioelectric Impedance Spectroscopy (BIS) can also be used.

Investigators postulate that it is possible to estimate GFR in the elderly from both SCr and LBM estimation from DXA. Proof of concept has already been made by others but until now, no specific formula for the elderly has been devised and properly validated.

Investigators'aim is thus to propose a new formula to predict GFR from both SCr and LBM (estimated from DXA) in the elderly. This formula will be elaborated from a first series of 100 patients and validated on a second series of 100 other patients.

ELIGIBILITY:
Inclusion criteria :

* age of 75 years of more
* origin from Western Europe or North Africa
* covered by social health insurance
* general health condition allowing transportation and ambulatory procedures during one day

Exclusion criteria :

* ascitis, oedema or third compartment
* fast change in body weight (more than 5% in less than one week)
* eGFR < 30 mL/min/1.73 m² (using MDRD formula)
* legal concerns: prisoners, guardianship, lack of health insurance, failure to consent
* intake of drugs that interfere with creatinine tubular secretion

  * cimetidine
  * trimethoprim
* intake of drugs that interfere with creatinine assay

  * calcium dobesilate
  * hydroxocobalamin
  * N-ethylglycine
  * phenindione
  * lidocaine
* inability to lie during 10 minutes without moving
* patients who are bedridden, hemiplegic or highly dependent on others
* any health condition that, in the investigator's opinion, could rapidly (< 1 week) vary the extracellular volume or GFR (these is voluntarily left open to the investigator because it is hardly possible to make an exhaustive list here)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-11-03 (Actual); Primary Completion 2022-11-02 (Estimated); Study Completion 2022-11-02 (Estimated)

PRIMARY OUTCOMES:
SCr and LBM estimated from DXA | Each participant is followed for one day.
  The formula that will be designed (using SCr and LBM estimated from DXA) from the first 100 patient data, will match measured GFR (as given by 51Cr-EDTA clearance) with less than 10 mL/min/1.73 m² absolute error in more than 90% of the other 100 patients.

SECONDARY OUTCOMES:
SCr and lean body mass ( by DXA) | Each participant is followed for one day.
  Detection of patient with impaired renal function by measuring SCr and lean body mass by DXA better than with existing formulas.
SCr and lean body mass (by BIS) | Each participant is followed for one day.
  A formula using SCr and measurement of lean body mass by bioelectric impedance spectrometry that will match measured GFR (as given by 51Cr-EDTA clearance) with less than 10 mL/min/1.73 m² absolute error in more than 90% of the other 100 patients.
SCr and morphological parameters | Each participant is followed for one day.
  A formula using SCr and measurement of morphological parameters (thigh perimeter, leg perimeter, arm perimeter) that will match measured GFR (as given by 51Cr-EDTA clearance) with less than 10 mL/min/1.73 m² absolute error in more than 90% of the other 10
Accuracy of new formulae | Each participant is followed for one day.
  The new formulae outperform eGFR (Cockcroft and Gault, MDRD and CKD-EPI formulae) for the following criteria: better accuracy (smaller bias) according to Bland and Altman
Precision of new formulae | Each participant is followed for one day.
  The new formulae outperform eGFR (Cockcroft and Gault, MDRD and CKD-EPI formulae) for the following criteria: better precision (smaller SD of difference) according to Bland and Altman.
Sensitivity of new formulae | Each participant is followed for one day.
  The new formulae outperform eGFR (Cockcroft and Gault, MDRD and CKD-EPI formulae) for the following criteria: sensitivity to detect GFR < 60 mL/min/1.73 m²
Specificity of new formulae | Each participant is followed for one day.
  The new formulae outperform eGFR (Cockcroft and Gault, MDRD and CKD-EPI formulae) for the following criteria: specificity to detect GFR < 60 mL/min/1.73 m²

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France